CLINICAL TRIAL: NCT00604799
Title: Evaluation of the Medtronic Vascular Talent Thoracic Stent Graft System for the Treatment of Thoracic Aortic Aneurysms
Brief Title: VALOR: The Talent Thoracic Stent Graft System Clinical Study
Acronym: VALOR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Investigational Plan #031
Record Dates: First submitted 2007-12-21; First posted 2008-01-30 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Thoracic Aortic Aneurysms
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Test (Enrollment Completed) (Active Comparator): Patients diagnosed with a TAA of degenerative etiology that are considered candidates for open surgical repair whom are low to moderate risk (0, 1, & 2) per the modified SVS/AAVS criteria who meet inclusion/exclusion criteria. The aneurysm must be at least 20 mm distal to the left common carotid artery & 20 mm proximal to the origin of the celiac artery.
  Interventions: Device: Talent Thoracic Stent Graft
- Registry (Enrollment Completed) (Other): Surgical candidates of low to moderate risk (SVS 0, 1, 2) that meet the Registry Inclusion/Exclusion criteria.
  Interventions: Device: Talent Thoracic Stent Graft
- High Risk (Enrollment Completed) (Other): Patients that meet one or more of the following:
  * High Risk (SVS 3)
  * Non-surgical candidates not associated with SVS scoring
  * Traumatic thoracic injuries
  Interventions: Device: Talent Thoracic Stent Graft
- Talent Captivia (Recruiting) (Other): Patients diagnosed with a TAA of degenerative etiology that are considered candidates for open surgical repair who meet inclusion/exclusion criteria.
  Interventions: Device: Talent Thoracic Stent Graft

INTERVENTIONS:
Device: Talent Thoracic Stent Graft — TEVAR

SUMMARY:
A Descending Thoracic Aneurysm is a bulge in the aorta. The aorta is a large blood vessel that carries blood away from your heart to organs in the rest of your body. Your aneurysm is caused by a weakening in the artery wall. If left untreated, this bulge may continue to grow larger and may ultimately rupture (break open) or extend in size to seriously affect other major arteries in the area. In this Research Study a device will be placed inside your aorta to block the weakened part of the artery wall from the circulatory system. Information will be collected on the performance for the device for 5 years.

ELIGIBILITY:
Talent Captivia Inclusion Criteria

1. Patient is at least 18 years of age.
2. Patient is a surgical or non-surgical candidate
3. Patient has a:

   1. Fusiform focal TAA AND / OR
   2. Focal saccular TAA or penetrating atherosclerotic ulcer.
4. Subject's anatomy must meet all of the following anatomical criteria:

   1. iliac/femoral access vessel morphology that is compatible with vascular access techniques, devices, and/or accessories
   2. non-aneurysmal aortic diameter in the range of 18-42mm; and
   3. non-aneurysmal aortic proximal and distal neck lengths =/>20mm
5. Thoracic aortic lesion is confirmed, at a minimum, by diagnostic contrast enhanced computerized tomography (CTA) with optional 3-D reconstruction, and/or contrast enhanced Magnetic Resonance Angiogram (MRA) obtained within the previous three (3) months prior to the implant procedure.
6. Subject or subject's legal representative understands and has signed an Informed Consent approved by the Sponsor and by the IRB for this study.
7. Patient must be able and willing to undergo follow-up imaging and examinations postoperatively up to 6 months.

Talent Captivia Exclusion Criteria

1. Planned placement of the COVERED (top edge of fabric) portion of the stent graft requires implant to occur in zones 0 or 1
2. Pregnant female
3. Patient has a connective tissue disease (e.g Marfan's syndrome, medial degeneration).
4. Patient has a mycotic aneurysm or is suspected of having systemic infection.
5. Patient has a history of bleeding diathesis, coagulopathy, or refuses blood transfusions.
6. Patient is currently participating in an investigational drug or device clinical trial that would interfere with the Talent Captivia protocol endpoints or follow-up.
7. The patient has known allergy or intolerance to the device components.
8. The patient has a known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment.
9. The patient has another medical condition, which may cause them to be non-compliant with the protocol, confound the data interpretation, or limited life expectancy of less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2003-07; Primary Completion 2006-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: proportion of patients in the Test Group who have successful aneurysm treatment at the 12-month follow-up visit. | 12 months
Primary Safety Endpoint: rate of "all cause" mortality of TAA repair with the Talent Thoracic Stent Graft against the literature control for open surgical repair within 1 year of follow-up. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kaye, MD, Principal Investigator — Physician's Regional Medical Center; Phillip Allmendinger, MD, Principal Investigator — Hartford Hospital; Mark Bates, MD, Principal Investigator — CAMC Health System; Daniel Benckart, MD, Principal Investigator — West Penn Allegheny Health System; Paul Bove, MD, Principal Investigator — Corewell Health East; Thomas Bower, MD, Principal Investigator — Mayo Clinic; Alfio Carroccio, MD, Principal Investigator — Mt. Sinai School of Medicine; Neal Cayne, MD, Principal Investigator — NYU Vascular Associates; Frank Criado, MD, Principal Investigator — Union Memorial Hospital; Alan Matsumoto, MD, Principal Investigator — University of Virginia; Mark Eskandari, MD, Principal Investigator — Northwestern Memorial Hospital; Ronald Fairman, MD, Principal Investigator — University of Pennsylvania; Mark Farber, MD, Principal Investigator — University of North Carolina; James McKinsey, MD, Principal Investigator — New York Presbyterian (Columbia & Cornell); Mark Fillinger, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center; H. Edward Garrett, MD, Principal Investigator — Baptist Memorial Hospital; Marc Glickman, MD, Principal Investigator — Sentar Norfolk General; Kim Hodgson, MD, Principal Investigator — Memorial Medical Center; Matthew Jung, MD, Principal Investigator — Surgical Care Associates; Barry Katzen, MD, Principal Investigator — Baptist Health South Florida; Zvonimir Krajcer, MD, Principal Investigator — St. Luke's Episcopal Hospital-Houston; Christopher Kwolek, MD, Principal Investigator — Massachusetts General Hospital; Lowell Satler, MD, Principal Investigator — Medstar Health Research Institute; Anthony Lee, MD, Principal Investigator — University of Florida; Alan Lumsden, MD, Principal Investigator — Baylor College of Medicine; Sean Lyden, MD, Principal Investigator — Cleveland Clinic Foundation-Ohio; Richard McCann, MD, Principal Investigator — Duke University; Manish Mehta, MD, Principal Investigator — Vascular Group, PLLC; Mark Mewissen, MD, Principal Investigator — St. Luke's Vascular Center; Takao Ohki, MD, Principal Investigator — Montefiore Medical Center; Venkatesh Ramaiah, MD, Principal Investigator — Arizona Heart Institute; Robert Rhee, MD, Principal Investigator — Shadyside Hospital-UPMC; Timothy Roush, MD, Principal Investigator — Carolinas Medical Center; Gregoria Sicard, MD, Principal Investigator — Washington University School of Medicine; Cary Stowe, MD, Principal Investigator — AdventHealth; Jim Swischuk, MD, Principal Investigator — Saint Francis Hospital; Michael Tuchek, MD, Principal Investigator — Loyola University; Rodney White, MD, Principal Investigator — Harbor UCLA; David Williams, MD, Principal Investigator — University of Michigan; Christopher Zarins, MD, Principal Investigator — Stanford University
Locations (1):
- University of Pennsylvania Hospital, Philadelphia, Pennsylvania, United States